CLINICAL TRIAL: NCT04053556
Title: Evaluation on the Effect on Cognition and Emotional Exhaustion With a Change of Long Night Shift System Versus Reduced Night Shift in Residents of Internal Medicine
Brief Title: Cognitive Performance After a Night Shift in Internal Medicine Residents
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Other Study IDs: 2489
Record Dates: First submitted 2016-10-26; First posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Sleep Deprivation; Burnout, Professional; Cognition Disorders
Keywords: sleep deprivation; internal medicine residency; on call; cognitive impairment; burn out; safety; depression
MeSH Terms: conditions — Sleep Deprivation; Burnout, Professional; Cognition Disorders; Cognitive Dysfunction; Burnout, Psychological; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A quasi-experimental design where internal medicine residents in a high complexity hospital were assessed after a 24-hour shift for cognitive impairment by a trained neurologist.

DETAILED DESCRIPTION:
The investigators conducted a cross sectional study during the 2014-2016 period in a high complexity school hospital in Buenos Aires. Second and third year Internal Medicine residents who consented to participate were included.

A neurologist conducted a cognitive evaluation to the residents who had done 24 hours shifts (with sleep deprivation) within 6 hours of its end.

Auditory memory deficit was evaluated (PASAT - Paced Auditory Serial Addition Test), verbal fluency (FAS), direct and indirect Digit-Span, Rey auditory verbal learning test (RAVLT) and Continuous Performance Test 2 (CPT2).

Results were presented as means of standardized scores (z score) with their interquartile range (IQR).

ELIGIBILITY:
Inclusion Criteria:

* Internal Medicine residents on the second or third year of formation.

Exclusion Criteria:

* Denial to participate in the study or to the informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Internal Medicine residents in formation who were on the second or third year of the Internal Medicine residency of the Italian Hospital of Buenos Aires who work 24 hours shifts and whose work day continues to a maximum of 36 total hours and who consented to the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Neurological evaluation using Paced Auditory Serial Addition Test (PASAT) | Immediately after a 24 hours on call period, wth a maximum delay of 6 hours after night shift end.
  Post on-call cognition assessment
Burn Out | through study completion, an average of one year
  Maslach questionaire filled by participant
Conners Continuous Performance Test 2 (CPT) | Immediately after a 24 hours on call period, wth a maximum delay of 6 hours after night shift end.
  Post on-call attention test
Rey auditory verbal learning test (RAVLT) | Immediately after a 24 hours on call period, wth a maximum delay of 6 hours after night shift end.
  Post on-call cognition assessment
F-A-S test | Immediately after a 24 hours on call period, wth a maximum delay of 6 hours after night shift end.
  Post on-call verbal fluency
Direct and indirect digit span | Immediately after a 24 hours on call period, wth a maximum delay of 6 hours after night shift end.
  Post on-call short-term verbal memory

SECONDARY OUTCOMES:
Depression | through study completion, an average of one year
  Questionaire filled by participant

CONTACTS AND LOCATIONS:
Overall Officials: Diego H Giunta, MD, Study Chair — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Peron 4190, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No